CLINICAL TRIAL: NCT05418010
Title: AttackMS: Natalizumab for the Treatment of People With Inflammatory Demyelination Suggestive of Multiple Sclerosis, or Definite Multiple Sclerosis, at First Presentation
Brief Title: Natalizumab for the Treatment of People With Inflammatory Demyelination Suggestive of Multiple Sclerosis, or Definite Multiple Sclerosis, at First Presentation (AttackMS)
Acronym: AttackMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Biogen (Industry); UCL Queen Square Institute of Neurology (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1003822; 2021-002255-11 (EudraCT Number)
Record Dates: First submitted 2022-02-17; First posted 2022-06-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome of Demyelination
Keywords: Multiple Sclerosis; Magnetic Resonance Imaging (MRI); Neurofilament light chain; Demyelinating Diseases; Immunologic Factors; Immune System Diseases; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Tyruko
MeSH Terms: conditions — Multiple Sclerosis; Charcot-Marie-Tooth disease, Type 1F; Demyelinating Diseases; Immune System Diseases; Autoimmune Diseases; Autoimmune Diseases of the Nervous System | interventions — Natalizumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled efficacy trial of hyperacute disease modifying treatment using Tyruko® in people with a first manifestation of central nervous system inflammatory demyelination.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tyruko® 300mg (Active Comparator): Tyruko® 300mg, administered via intravenous infusion in a 4 week cycle, for a total of 6 cycles
  Interventions: Drug: Tyruko Injectable Product
- Placebo (Placebo Comparator): Placebo, administered via intravenous infusion in a 4 week cycle, for 3 cycles, followed by Tyruko® 300mg, administered via intravenous infusion for a total of 3 cycles
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tyruko Injectable Product — Tyruko® is indicated as single disease modifying therapy in adults with highly active relapsing remitting multiple sclerosis. Tyruko® 300mg concentrate for solution for infusion and matching placebo are collectively referred to as IMP when detailing to blinded trial procedures. Tyruko® 300mg will be colourless, clear to slightly opalescent solution.
  Other Names: Natalizumab
  Arms: Tyruko® 300mg
Drug: Placebo — Placebo is colourless, clear to slightly opalescent liquid. The formulation of the is the same as that of commercial Tyruko® minus the active ingredient. Placebo is in the same containers/vials as Tyruko®.
  Arms: Placebo

SUMMARY:
Multiple Sclerosis (MS) is a chronic inflammatory & degenerative disease of the central nervous system (CNS) Recent data from the MS Base registry demonstrated an average delay of 152 - 215 days between first presentation and the diagnosis of MS, and more than one year until Disease Modifying Treatment (DMT) begins.

Evidence suggests that shutting down inflammation using highly effective DMTs early after diagnosis leads to better long term clinical outcomes The AttackMS trial will test the effect of starting a highly-effective DMT licensed for MS, Tyruko® (Natalizumab 300mg), within a short time - 14 days - after symptom onset.

DETAILED DESCRIPTION:
MS is a disease of the central nervous system affecting over 130,000 people in the UK and more than 2.8 million worldwide. Left untreated, MS leads to chronic disability in the large majority of cases.

CIS is a common first manifestation of MS: There is a more than 80% chance of MS in somebody presenting with CIS provided one or more "lesions" characteristic of inflammatory demyelination can be detected on a magnetic resonance imaging (MRI) of the brain. The presence of at least two such lesions is an inclusion criterion for this study. Inflammatory demyelination is the process by which cells of your body's own immune system attack the insulation sheath (= myelin) of nerve fibres (= axons) in the central nervous system.

Once a diagnosis of MS has been confirmed, many people with this disease will be eligible for what is called "disease-modifying treatment" (DMT) on the NHS. Such treatment targets the immune cells that are involved in the inflammatory attack against the myelin sheaths and nerve fibres. However, while in a small number of cases, a diagnosis of MS can be made instantaneously it regularly takes week, months and, sometimes even longer, to fulfil the formal diagnostic criteria of MS. This diagnostic delay inevitably leads to delays in starting disease-modifying treatment.

Using a trial concept geared towards rapid assessment of eligibility, and a disease-modifying treatment that is both highly effective and generally well tolerated in people with MS, AttackMS will test whether:

(i) It is feasible to recruit participants with a diagnosis of CIS at high risk of MS, or definite MS, at first presentation for treatment within 14 days of symptom onset and (ii) Such early treatment improves myelin repair at 3 months, as measured using a special MRI technology called magnetisation transfer ratio (MTR).

Natalizumab (Tyruko®) is a medication currently approved by the Medicines and Healthcare products Regulatory Agency (MHRA) as a disease-modifying treatment for adults with rapidly evolving severe (RES) relapsing MS. We are looking to test safety and efficacy of treatment with Tyruko® 300mg, given through a needle in a vein (intravenous infusion), over 20 weeks and to advance mechanistic understanding in treating people with first presentation of CIS or MS.

AttackMS will test the effect of starting a highly-effective DMT licensed for MS, Tyruko®, within a short time - 14 days - after symptom onset. The main objective is to test Tyruko®, given intravenously every 4 weeks over 20 weeks, for safety, efficacy, and to advance the mechanistic understanding of the earliest events in inflammatory demyelination/MS.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent.
2. Age 18-55 years
3. Participant with CIS or MS at first presentation.
4. Participants show two or more lesions on T2 weighted MRI suggestive of demyelination.
5. Participant is willing and able to comply with clinical visits and procedures outlined in the study protocol.

Exclusion Criteria:

1. Hypersensitivity to Tyruko® or to any of the following excipients:

   * Histidine
   * Histidine monohydrochloride
   * Sodium chloride
   * Polysorbate 80 (E433)
   * Water for injections
2. Evidence of multiple chronic demyelinating lesions on MRI without signs of recent activity.
3. Participants with increased risk for opportunistic infections, including immunocompromised participants (those currently receiving immunosuppressive therapies or those immunocompromised by prior therapies).
4. Combination with other Disease Modifying Treatments..
5. Known active malignancies, except for participants with cutaneous basal cell carcinoma.
6. Implants such as pacemaker, aneurysm clip in the brain and MRI-incompatible prosthetic heart valves.
7. Significant comorbidities such as cardiac failure, renal failure, uncontrolled diabetes and uncontrolled hypercholesterolemia.
8. History of stroke, thrombosis and/or myocardial infarction.
9. Any other infection deemed, in the assessment of the PI or sub-investigator, clinically significant.
10. Claustrophobia
11. Pregnancy or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To establish whether there is efficacy superiority of Natalizumab (Tyruko®) over placebo at 12 weeks in facilitating remyelination of previously demyelinated CNS lesions, as measured by MRI lesion magnetization transfer ratio (MTR). | 12 weeks
  Mean magnetisation transfer ratio (MTR) change in FLAIR-hyper-intense lesions at 12 weeks compared to baseline

SECONDARY OUTCOMES:
To establish whether there is a difference between participants receiving Natalizumab (Tyruko®) or placebo at 24 weeks in P100 latency measured using visually evoked potentials (VEP). | 0 and 24 weeks
  P100 latency in each eye at week 24 compared to baseline. Inter-ocular P100 latency difference at week 24 compared to baseline.
To establish whether there is a difference between participants receiving Natalizumab (Tyruko®) or placebo at 24 weeks in number and occurrence of adverse events. | 24 weeks
To establish whether there is a difference between participants receiving Natalizumab (Tyruko®) or placebo at 24 weeks in facilitating remyelination of previously demyelinated CNS lesions using Magnetisation transfer ratio (MTR). | 0, 12 and/or 24 weeks
To establish whether there is a difference between participants receiving Natalizumab (Tyruko®) or placebo at 24 weeks in protecting limb function. | 24 weeks
  Serum-neurofilament light chain levels (SNfL) at week 24 compared to baseline. Expanded Disability Status Scale (EDSS) at week 24 compared to baseline. SDMT (Symbol Digit Modalities Test) score at week 24 compared to baseline. Lower Limb Function: The T25-FW (Timed 25 Foot Walk) will be collected in all pwMS. able to walk the required distance at week 24 compared to baseline.
  9-HPT (Nine Hole Peg Test) at week 24 compared to baseline. NFI-MS (Neurological Fatigue Index-MS) score at week 24 compared to baseline 24 weeks.
To establish whether there is a difference between participants receiving Natalizumab (Tyruko®) or placebo at 24 weeks in Retinal nerve fibre layer ganglion cell + inner plexiform (GCIP) layer thickness measured using optical coherence tomography (OCT). | O and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schmierer, Principal Investigator — Queen Mary University of London; Liqun Zhang, Principal Investigator — St George's University Hospital NHS Foundation Trusts; Victoria Singh-Curry, Principal Investigator — Chelsea and Westminster Hospital Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal London Hospital, London
  - St George's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
IPD data collected on the trial will be uploaded to the Pragmatic Clinical Trials Unit Safehaven and linked using pseudoanonymised participant IDs. Any further sharing of participant data to other researchers will be fully anonymised as specified at the time of participant consent.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: AttackMS Abstract — https://jnnp.bmj.com/content/jnnp/93/9/e2.108.full.pdf
- See also: CI Interview: AttackMS assessing the feasibility of multiple sclerosis treatment within 14 days of presentation — https://www.youtube.com/watch?v=uhkHZqXRIpM
- See also: Multiple Sclerosis Academy Webinar on AttackMS — https://neurologyacademy.org/events/webinar/what-does-treating-ms-early-mean-in-clinical-practice

DOCUMENTS (1):
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT05418010/ICF_001.pdf